CLINICAL TRIAL: NCT01922661
Title: Single Ascending-dose Study of the Safety, Tolerability, and Pharmacokinetics of REGN1908-1909 in Allergic, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R1908-HV-1240
Record Dates: First submitted 2013-08-02; First posted 2013-08-14 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Dose 1 of REGN1908-1909 or placebo
  Interventions: Drug: REGN1908-1909; Other: placebo
- Cohort 2 (Experimental): Dose 2 of REGN1908-1909 or placebo
  Interventions: Drug: REGN1908-1909; Other: placebo
- Cohort 3 (Experimental): Dose 3 of REGN1908-1909 or placebo
  Interventions: Drug: REGN1908-1909; Other: placebo

INTERVENTIONS:
Drug: REGN1908-1909
Other: placebo

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of single ascending doses of subcutaneously (SC) administered REGN1908-1909 in allergic, adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between the ages of 18 and 55
2. Positive allergen skin prick test
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Exclusion Criteria:

1. Persistent, chronic, or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the screening visit
2. Any clinically significant (determined at the investigator's discretion) abnormalities observed during the screening physical examination
3. Onset of a new exercise routine or major change to a previous exercise routine within 4 weeks prior to the screening visit. Patients must be willing to maintain a similar level of exercise for the duration of the study and to refrain from unusually strenuous exercise for the duration of the trial
4. Hospitalization for any reason within 60 days prior to the screening visit
5. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer) of the investigational drug prior to the screening visit
6. Any medical or psychiatric condition that in the opinion of the investigator or Regeneron, would place the patient at risk, interfere with participation in the study or interfere with the interpretation of study results

The information listed above is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial and not all inclusion/ exclusion criteria are listed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety | day 1 to day 113
  The primary endpoint is to assess treatment-emergent adverse events (TEAEs) from day 1 through day 113 (end of study).

SECONDARY OUTCOMES:
Serum concentration | day 1 to day 113
  The secondary endpoint is serum concentrations of REGN1908-1909 over time.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Overland Park, Kansas
  - Baltimore, Maryland

REFERENCES:
- [Derived] Kamal MA, Dingman R, Wang CQ, Lai CH, Rajadhyaksha M, DeVeaux M, Orengo JM, Radin A, Davis JD. REGN1908-1909 monoclonal antibodies block Fel d 1 in cat allergic subjects: Translational pharmacokinetics and pharmacodynamics. Clin Transl Sci. 2021 Nov;14(6):2440-2449. doi: 10.1111/cts.13112. Epub 2021 Aug 26. PMID 34437752